CLINICAL TRIAL: NCT04694846
Title: Feasibility of the Enhanced Tobacco Intervention Protocol (ETIP) to Reduce Smoking and Potentially Alter the Tumor Microenvironment of Head and Neck Squamous Cell Carcinoma and Non-Small Cell Lung Cancer
Brief Title: Effectiveness of an Enhanced Tobacco Intervention Protocol Compared to Standard Treatment in Helping Head and Neck and Lung Cancer Patients Starting Treatment to Reduce Cigarette Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19D.866; JT 14301 (Other: JeffTrial Number)
Record Dates: First submitted 2020-03-16; First posted 2021-01-05 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Lung Non-Small Cell Carcinoma; Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck | interventions — Nicotine Replacement Therapy; Bupropion; Varenicline; Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (ETIP) (Experimental): Patients receive nicotine replacement therapy via trans-dermal patch, gum, nasal spray, inhaler or lozenges for 12 weeks in the absence of unacceptable toxicity. Patients also receive bupropion PO QD BID or varenicline PO QD and BID for 24 weeks in the absence of unacceptable toxicity. Patients undergo 3 cessation counseling sessions in person, via telehealth or phone within 7 days of enrollment into study, 1 week after established quit date and 3 weeks after establishing quit date.
  Interventions: Drug: Nicotine Replacement; Drug: Bupropion Hydrochloride Controlled-release; Drug: Varenicline; Other: Tobacco Cessation Counseling; Other: Questionnaire Administration; Other: Quality of Life Assessment
- Arm II SOC (Active Comparator): Participants randomly assigned to the standard treatment (ST) group will receive an in-office smoking cessation recommendation by the physician and referral to a quit line.
  Interventions: Other: Questionnaire Administration; Other: Quality of Life Assessment; Other: Best Practice

INTERVENTIONS:
Drug: Nicotine Replacement — Given NRT via trans-dermal patch, gum, nasal spray, inhaler or lozenges
  Other Names: nicotine replacement therapy, Nicotine Replacement Therapy, NRT
  Arms: Arm I (ETIP)
Drug: Bupropion Hydrochloride Controlled-release — Given PO
  Other Names: Bupropion HCl Controlled-release, Bupropion HCl Extended Release, Bupropion Hydrochloride Extended-Release, Forfivo XL, Wellbutrin SR, Wellbutrin XL, Zyban, Zyban
  Arms: Arm I (ETIP)
Drug: Varenicline — Given PO
  Other Names: 249296-44-4, 7,8,9,10-tetrahydro-6,10-methano-6H-pyrazino(2,3-h)(3)benzazepine (2R,3R)-2,3-dihydroxybutqanedioate, Champix, Chantix, CP-526555, VARENICLINE
  Arms: Arm I (ETIP)
Other: Tobacco Cessation Counseling — Receive counseling
  Arms: Arm I (ETIP)
Other: Questionnaire Administration — Ancillary studies
Other: Quality of Life Assessment — Ancillary studies
Other: Best Practice — Receive standard treatment
  Other Names: best practice, standard of care, standard of care, standard therapy
  Arms: Arm II SOC

SUMMARY:
This trial studies how well an enhanced tobacco intervention protocol (ETIP) works compared to standard treatment in helping head and neck and lung cancer patients starting treatment to reduce cigarette use. ETIP is an evidence-based tobacco cessation program including specialized one-to-one and telehealth counseling, drug therapy, nicotine replacement therapy, and frequent patient follow up. ETIP may help reduce smoking and improve cessation in patients with head and neck squamous cell cancer or non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility of implementing a transdisciplinary ETIP using enrollment data and adherence to the intervention.

SECONDARY OBJECTIVE:

I. To compare smoking reduction, physiologic parameters and patient reported measures among patients in two tobacco treatment groups (ETIP and standard treatment [ST]).

TERTIARY OBJECTIVE:

I. To determine patient interest in wellness practices as a means to alter behavior and facilitate tobacco cessation.

EXPLORATORY OBJECTIVES:

I. To analyze the genetic profile, serum and tissue exosomal signatures, and immune cell profiles of both human papilloma virus (HPV) positive and negative tumor samples in patients who are never smokers, former smokers, and current smokers.

II. Compare these parameters in patients who underwent ETIP versus standard therapy.

III. To gather correlative data regarding the effects of tobacco smoke on the expression of biomarkers and the tumor microenvironment.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (ETIP): Patients receive nicotine replacement therapy via trans-dermal patch, gum, nasal spray, inhaler or lozenges for 12 weeks in the absence of unacceptable toxicity. Patients also receive bupropion orally (PO) once daily (QD) and twice daily (BID) or varenicline PO QD and BID for 24 weeks in the absence of unacceptable toxicity. Patients undergo 3 cessation counseling sessions in person, via telehealth or phone within 7 days of enrollment into study, 1 week after established quit date and 3 weeks after establishing quit date.

ARM II (ST): Patients receive standard treatment consisting of an in-office smoking cessation recommendation by the physician and referral to a quit line.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed written informed consent document
* New patients opting to receive cancer care at Thomas Jefferson University Hospital (TJUH) or Methodist with suspected or newly diagnosed head and neck squamous cell carcinoma (HNSCC) or non-small cell carcinoma of the lung
* Must have a life expectancy of at least 6 months as judged by the treating physician
* Willing to discuss changing their smoking behavior
* Patients have smoked > 100 cigarettes in their lifetime and have smoked within the last 30 days
* Subjects must read and speak fluent English

Exclusion Criteria:

* Patients with psychiatric disorders with indications of current uncontrolled illness, or patients currently being treated on psychiatric medications
* Patients with expected survival of less than 6 months or other medical illness that would prevent participation as determined by the treating clinician
* Patients not fluent in English will be excluded, as the counselling component of the intervention is only available in English
* Pregnant or breastfeeding women
* Severe swallowing disorders or other illness that would impede a patient's ability to swallow medications in pill form
* Patients with impaired judgement or those unable to provide informed consent
* Contraindications to nicotine replacement therapy:

  * All free flap patients: Nicotine replacement therapy (NRT) and tobacco products must not be used by these patients for at least 2 weeks before and 2 weeks after free flap surgery. For planned procedures involving face and breast, tobacco and NRT use should be avoided 4 weeks before and 4 weeks after surgery
  * Patients in the immediate (within 2 weeks) post myocardial infarction period or who have serious arrhythmias or unstable angina pectoris
  * Patient who are hemodynamically or electrically unstable or have had orthopedic surgery or a serious fracture(s) within the past 6 weeks
  * Patients with known allergy or hypersensitivity to NRT, or severe skin reactions like Steven's Johnson syndrome
* Contraindications to bupropion or varenicline:

  * Pre-existing seizure disorder or conditions that increase the risk of seizures (e.g., severe head trauma, arteriovenous malformation, central nervous system (CNS) tumor (e.g., brain tumor or intracranial mass), CNS infection, severe stroke, anorexia nervosa, bulimia nervosa
  * Patients undergoing abrupt discontinuation of alcohol, benzodiazepines, barbiturates, and antiepileptic drugs
  * Concomitant use of anti-depressants
  * Patients with known allergy or hypersensitivity to bupropion or varenicline, or severe skin reactions like Steven's Johnson syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Reduction in daily number of cigarettes smoked by at least 50% compared to baseline at months 1 and 6 | Up to 6 months
  This will be biochemically verified by any reductions in minor tobacco alkaloid (anabasine/anatabine) concentrations in the urine compared to baseline

SECONDARY OUTCOMES:
Cigarette abstinence at 1 and 6 months, as reported by patients | Up to 6 months
  Subjects with missing data will be counted as smokers
Proportion of patients having urine anabasine/anatabine levels of less than 2ng/ml | Up to 6 months
  Participants will be asked to provide a urine sample for biochemical verification of smoking status with urine anatabine/anabasine testing at baseline, 1 and 6 months. We consider urine anabasine/anatabine less than or equal to 2 ng/ml to be evidence of abstinence. Participant failure to provide a sample will be interpreted as biochemical evidence of smoking.

OTHER OUTCOMES:
Interest expressed in wellness practices | Up to 6 months
  Descriptive statistics (means and standard deviations for continuous variable and frequencies for categorical variables) will be used to summarize interest in wellness programs.
Types of wellness practices patients prefer | Up to 6 months
Likelihood of patient participation | Up to 6 months
Modes of intervention delivery | Up to 6 months
  Descriptive statistics (means and standard deviations for continuous variable and frequencies for categorical variables) will be used to summarize referred time and method of program delivery.
Biomarker analysis | Up to 6 months
  Immunohistochemistry (IHC) analysis will be done on all patient tissue samples at the initial visit. Additionally, serum blood samples will be collected from all patients. Serum c-reactive protein (CRP) and lipid levels will be tested at various time points in the study to account for changes in inflammatory marker expression. Peripheral blood assays, including Luminex, will be used to quantify immune mediators including expression of interferon (IFN)-gamma, IL-2, and IL-10 among other analytes.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sidney Kimmel Cancer Center at Thomas Jefferson Univeristy, Philadelphia, Pennsylvania
  - Jefferson Health, Methodist Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No